CLINICAL TRIAL: NCT06038396
Title: A Phase I/II Clinical Study to Evaluate the Safety and Efficacy of RC118 in Combination with Toripalimab / RC148 for Patients with Claudin 18.2-Positive, Locally Advanced Unresectable or Metastatic Malignant Solid Tumors
Brief Title: A Study of RC118 Plus Toripalimab / RC148 in Patients with Locally Advanced Unresectable or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RC118-C002
Record Dates: First submitted 2023-09-01; First posted 2023-09-14 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-09

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — Injections; toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part A-RC118 plus Toripalimab (Experimental): Participants receive RC118- ADC(dose A or dose B) Q2W and Toripalimab (fixed dose) Q3W
  Interventions: Drug: RC118; Drug: Toripalimab
- Part B-RC118 plus Toripalimab / RC148 (Experimental): Referring to the results of the Part A, an extension cohort using RC118 plus Toripalimab /RC148 will be established.
  Interventions: Drug: RC118; Drug: Toripalimab; Drug: RC148

INTERVENTIONS:
Drug: RC118 — Dose A or dose B, Q2W
  Other Names: RC118 for injection
Drug: Toripalimab — Fixed dose, Q3W
  Other Names: Toripalimab injection; JS001
Drug: RC148 — Fixed dose, Q3W Other Names: RC148 injection
  Arms: Part B-RC118 plus Toripalimab / RC148

SUMMARY:
This is an open, multi-center, dose escalation and expansion phase I/II study. The Phase I study will explore the tolerability and safety of RC118 in combination with Toripalimab for the treatment of patients with Claudin 18.2-positive, locally advanced unresectable or metastatic malignant solid tumors, and to establish the maximum tolerated dose (MTD) and the recommended dose in phase II clinical trials (RP2D); The Phase II study will evaluate the efficacy and safety of RC118 in combination with Toripalimab or RC148 in patients with locally advanced or metastatic Gastric cancer/Gastro-esophageal junction cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to participate in the study voluntarily and willing to provide written informed consent.
2. male or female 18 ≤ age ≤ 75 years old.
3. Must have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
4. The expected survival ≥12 weeks.
5. Enrollment of subjects with locally advanced or metastatic gastric adenocarcinoma/adenocarcinoma of the gastroesophageal junction who have a histologically confirmed diagnosis and have failed standard therapy.
6. Subjects who received ≤2 prior systemic therapies.
7. Subjects agree to provide tumor tissue specimens for Claudin 18.2 and PD-L1 expression levels during the screening period. Samples should have moderate to high expression of Claudin 18.2 by membrane staining.
8. According to the RECIST v1.1, there is at least one measurable target lesion.
9. Sufficient heart, bone marrow, liver and kidney functions.
10. Fertile male or female subjects must agree to take effective contraceptive measures during the study period and for 6 months after the end of the last dose, such as double-barrier contraceptive methods(eg. condoms), oral or injectable contraceptives, intrauterine.

Exclusion Criteria:

1. Pregnant women, breastfeeding women or women with a positive blood pregnancy test result during the screening period (non-fertile women do not need to undergo a pregnancy test, such as women with a previous hysterectomy and/or bilateral oophorectomy or amenorrhea ≥12 months).
2. Subjects with active hepatitis B (HBsAg positivity and HBV DNA titre higher than the normal upper limit), active hepatitis C (HCVAb positivity and HCV RNA titre higher than the normal upper limit), and positive human immunodeficiency virus antibody (HIV-Ab) results during the screening period.
3. Subjects with a history of other acquired or congenital immunodeficiency diseases, or who have undergone organ or bone marrow transplantation.
4. Subjects who have previously received monoclonal antibody, double antibody targeting drugs, ADC, CAR-T and other therapeutic drugs targeting Claudin 18.2 or other ADCs with MMAE payload; or have participated in clinical trials and received investigational drugs within 4 weeks before the first dose.
5. Have vaccinated within 4 weeks prior to the first dose or plan to receive any live vaccine during the study.
6. Subjects are atallergic to the ingredients or excipients of the experimental drug.
7. Subjects who have received anti-tumor therapy (chemotherapy, radiotherapy, immunotherapy, or targeted therapy) within 4 weeks or less than 5 half-lives of the experimental drug prior to the start of the first dose; or who have received anti-tumor therapy with traditional Chinese medicine or immunomodulators within 2 weeks prior to the start of the first dose.
8. The toxicity of previous anti-tumor therapy has not returned to the level 0 or 1 as defined by NCI-CTCAE v5.0 (except for alopecia, pigmentation and other long-term toxicity ≤2 that cannot be recovered which was defined by investigators).
9. The clinical symptoms of pleural effusion, abdominal effusion, or pericardial effusion that requires drainage.
10. Active infection within 2 weeks prior to the first dose that requires systemic anti-inflammatory therapy.
11. Complicating other diseases that seriously endanger the safety of the subjects or affect the completion of the study, such as peptic ulcer, intestinal obstruction, intestinal paralysis, interstitial pneumonia, pulmonary fibrosis, renal failure and uncontrolled diabetes (Fasting blood glucose > 8.5 mmol/L, HbA1C ≥7.5%).
12. The tumor lesion has a bleeding tendency or has received blood transfusion treatment within 4 weeks prior to the first dose.
13. During the screening period, QTc interval >450 ms(male), QTc interval >470ms(female); previous family or personal history of long/short QT interval syndrome; A history of ventricular arrhythmia deemed clinically significant by the investigator, or currently receiving antiarrhythmic medication, or implantation of arrhythmia defibrillation device.
14. Previous myocardial infarction (within 6 months prior to the first dose), severe or unstable angina, coronary or peripheral artery bypass grafting, heart failure grade 3~4 defined by New York Heart Association (NYHA) and uncontrolled hypertension.
15. Experienced an arterial/venous thromboembolic event within 6 months prior to the study.
16. Active autoimmune disease that requires systemic treatment within 2 years prior to the study. Patients with vitiligo, psoriasis, alopecia or Grave's disease that not requires systemic treatment, hypothyroidism that only requires thyroid hormone replacement therapy, and type 1 diabetes only requires insulin replacement therapy may be included in the study.
17. Subjects with brain metastases and/or carcinomatous meningitis who have previously received related treatment may be considered for inclusion if their disease has been stable for at least 3 months, no imaging evidence of disease progression has been observed within 4 weeks prior to the first dose, all neurological symptoms have returned to baseline, and radiation, surgery, or steroid therapy has been discontinued at least 28 days prior to the first dose; cancerous meningitis should be excluded regardless of whether it is clinically stable.
18. Other malignant tumor within 5 years prior to the signature of informed consent.
19. Major surgery or interventional therapy was performed within 4 weeks prior to the first dose and did not fully recovered (except tumor biopsy and puncture).
20. For Phase II subjects:

    * Received an immune checkpoint inhibitor (anti-PD-1/PD-L1/CTLA-4 antibody) or other immune checkpoint inhibitor therapy within 28 days prior to the first treatment with the test drug;
    * Prior concurrent receipt of antitumor agents targeting VEGF/VEGFR and PD-1/PD-L1;
    * Experienced permanent discontinuation of immunotherapy due to toxicity of immune checkpoint inhibitor therapy prior to receiving administration of study drug;
    * Currently receiving anticoagulant medications (except for subjects on prophylactic doses of heparin).
21. A history of uncontrollable mental illness or subjects currently experiencing such conditions.
22. Subjects with poor compliance who are expected to be unable to complete the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-08-03 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Phase1: Dose limiting toxicity (DLT) | The first 3 weeks (21 days) after the start of dosing at each dose level
  Toxicity occurs within the DLT evaluation window (1-21 days after the first dose) that the investigator or sponsor believes to be reasonably associated with RC118 or Toripalimab according to NCI-CTCAE v5.0.
Phase1/2: Adverse events (AEs) | [Time Frame: 15 months]
  Incidence and severity of adverse events (AEs) and serious adverse events (SAEs), and clinically significant abnormal laboratory results.
Phase1: Maximum tolerated dose(MTD) | up to 12 months
  Maximum tolerated dose(MTD)
Phase1: Recommended Phase 2 Dose (RP2D) | up to 12 months
  Recommended Phase 2 Dose (RP2D)
Phase 2: Objective response rate (ORR) | 15 months
  The proportion of patients whose BOR is a confirmed CR or PR. Tumor response will be evaluated using RECIST v.1.1.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | 15 months
  The percentage of patients who have achieved an objective response of confirmed CR ,PR or SD as assessed by the investigator per RECIST v1.1)
Progression-free survival (PFS) | 15 months
  The time from first dose to disease progression(as assessed by investigators according to RECIST v1.1 criteria) (as measured by the first event).
Duration of Remission (DOR) | 15 months
  The time from first documentation of response (CR or PR) until the time of first documentation of disease progression or death.
Overall survival (OS) | 15 months
  The time from the date of the first dose of study treatment to the date of death.
Phase 1: Objective response rate (ORR) | 15 months
  The proportion of patients whose BOR is a confirmed CR or PR. Tumor response will be evaluated using RECIST v.1.1.
Peak and valley concentrations of RC118, total antibody, and free MMAE | 15 months
  Peak and valley concentrations of C118 binding antibody, total antibody, and free MMAE were observed.
RC118 immunogenicity: The incidence, time of onset, duration of patients with anti-drug-antibody (ADA) | 15 months
  RC118 immunogenicity: The incidence, time of onset, duration of patients with anti-drug-antibody (ADA)

CONTACTS AND LOCATIONS:
Overall Officials: Tianshu Liu, ph.D, Principal Investigator — Shanghai Zhongshan Hospital
Locations (18):
- China (18):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Gansu Wuwei Tumour Hospital, Wuwei, Gansu
  - Meizhou People's Hospital, Meizhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Nanyang Central Hospital, Nanyang, Henan
  - Xinyang Central Hospital, Xinyang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Bengbu Medical University, Bengbu, Shandong
  - Cancer Hospital of Shandong First Medical University, Jinan, Shandong
  - Changzhi People's Hospital, Changzhi, Shanxi
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - The Second People's Hospital of Neijiang, Neijiang, Sichuan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Zhongshan Hospital Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: No